CLINICAL TRIAL: NCT03046797
Title: Boussignac Valve and Fibroptic Intubation in Morbidly Obese Patients, Can it be a Solution?
Acronym: Obese-FOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Obese-FOB
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B group (Experimental): Mask ventilation will be continued and fiberoptic intubation will be performed from Boussignac valve opening by an experienced anesthetist.
  Interventions: Device: Fibroptic intubation through Boussignac valve opening
- C group (Active Comparator): mask ventilation will be terminated then fiberoptic intubation will be done by an experienced anesthetist.
  Interventions: Device: Classic Fibroptic intubation

INTERVENTIONS:
Device: Fibroptic intubation through Boussignac valve opening — After patients being put in HELP position to facilitate both ventilation and intubation, mask ventilation will be continued and FOB intubation will be performed from Boussignac valve opening.
  Arms: B group
Device: Classic Fibroptic intubation — After patients being put in HELP position to facilitate both ventilation and incubation, mask ventilation will be terminated then FOB intubation will be done by an experienced anesthetist.
  Arms: C group

SUMMARY:
In this study, fiberoptic intubation through Boussignac valve, while ventilation of morbidly obese patients is maintained through the ventilator, will be studied. Researchers suggest that the technique will allow more time for intubation trial rather than conventional techniques of intubation without ventilation. the Primary outcome will be the decrease of desaturation events during intubation. Secondary variables will include; stress response to intubation, the incidence of hypercapnia, hemodynamic response to intubation, successful intubation, the time required to intubation and operator satisfaction.

DETAILED DESCRIPTION:
All patients will be subjected to a thorough preoperative evaluation including clinical assessment, ECG, Echocardiography, pulmonary function tests and laboratory investigations (CBC, SGOT, SGPT, Albumin, Serum creatinine) and basal arterial blood gases. All patients will be pre-medicated with intravenous infusion of pantoprazole (40 mg) and metoclopramide (10 mg). After pre-oxygenation with 100% oxygen for 5 minutes, anesthesia will be induced using propofol (1-2 mg/kg) preceded by 60 mgs of lidocaine, and rocronium (0.12 mg/kg). Mask ventilation will be maintained while a Boussignac valve is attached between the Y-circuit and the face mask. After full relaxation is achieved (60 second after TOF response disappears), intubation attempt will commence.

Intubation technique:

Patients of both, patients will be put in HELP position to facilitate both ventilation and incubation

* In C group: mask ventilation will be terminated then FOB intubation will be done by experienced anesthist.
* In B group: Mask ventilation will be continued and FOB intubation will be performed from Boussignac valve opening.

Data collection:

Patient demographic data (Age, Weight, height, BMI, ASA status, coexisting diseases) will be collected. Hemodynamic parameters will be r5ecorded at the following points (Preoperative, basal, 1,2,3 minutes after starting intubation attempt).

Time to successful intubation will be documented in seconds (starting from passing of FOB through mouth opening till successful placement of the tube in the trachea). Also, time to glottis visualization and time to carina visualization will be recorded. Number of attempts will be also recorded where unsuccessful attempt will be defined as the need to withdraw FOB outside the patient's mouth (either due to failure to progress or need for ventilation). a desaturation event will be defined as SpO2 less than 94. Also, any procedure-related complication will be documented (hypertension, arrhythmia, spasm, bleeding) Statistical analysis G*power software version 3.1.9.2 was used for sample size calculation. We assumed that using Boussignac valve during FOB intubation can produce a 20% increase in the time to reach patients spo2 of 95% (180±20 sec in previous studies). It was found that 16 patients per was required to achieve a power of 90% with an alpha error of 0.05. additional 4 patients were added to compensate or dropouts making a total sample size of 40 patients.

Data will be collected and tabulated in excel sheet (Microsoft office, 2016). Statistical analysis will be performed using SPSS software version 20. Continuous data will be tested for normality of distribution and presented as mean±SD or median (interquartile range). Statistical differences between the studied groups will be assessed using appropriate statistical tests

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients (BMI above 40kg/m2) scheduled for elective surgery, with age between 20 to 45 years

Exclusion Criteria:

* unstable ischemic heart disease, uncontrolled systemic hypertension, previous history of difficult intubation and patients with basal oxygen saturation less than 94%

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
number of desaturation events | 3 minutes after the start of intubation attempt
  desaturation (spo2 less than 94) during fibroptic intubation of morbidly obese patients

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura university, Al Mansurah, Dkahleya
  - Gastroenterology center, Al Mansurah

IPD SHARING:
Plan to Share IPD: Undecided